CLINICAL TRIAL: NCT00075569
Title: SGN-00101 (HspE7) Immunotherapy Of CIN III
Brief Title: SGN-00101 Immunotherapy in Treating Patients With Grade III Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03-10-251; AECOM-0309225 (Other: Albert Einstein College of Medicine); NCI-5850 (Other Grant/Funding Number: National Cancer Institute)
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2006-01

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Parallel design

ARMS (2):
- 1 month follow-up (Active Comparator): 3 monthly subcutaneous vaccinations with 500 microg of HspE7 followed by monthly colposcopic follow-up for 1 month; followed by LEEP or cone biopsy
  Interventions: Biological: HspE7
- 2 month follow-up (Active Comparator): 3 monthly subcutaneous vaccinations with 500 microg of HspE7 followed by monthly colposcopic follow-up for 2 months; followed by LEEP or cone biopsy
  Interventions: Biological: HspE7

INTERVENTIONS:
Biological: HspE7 — 500 micrograms of SGN-00101 (HspE7, Nventa, San Diego, CA) is a novel therapeutic vaccine consisting of a fusion protein containing an M. bovis BCG heat shock protein (Hsp65) covalently linked to the entire sequence of HPV 16 E7.
  Other Names: SGN-00101

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of cancer or to treat early cancer. SGN-00101 may be effective in preventing the development of cervical cancer in patients who have cervical intraepithelial neoplasia.

PURPOSE: This phase II trial is studying how well SGN-00101 immunotherapy works in preventing cervical cancer in patients with grade III cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the rate of regression at 4-7 months in patients with grade III cervical intraepithelial neoplasia (CIN III) treated with SGN-00101 immunotherapy.
* Compare the rate of regression at 4-7 months with expected outcome in patients immunized with this vaccine.
* Determine the toxic effects and recovery from possible toxic effects of this vaccine in these patients.

Secondary

* Determine induction of cell-mediated immune responses against human papillomavirus (HPV) E7 peptides before and after treatment in patients immunized with this vaccine
* Correlate regression of disease with enhanced immunologic responses in patients immunized with this vaccine.
* Correlate seropositivity of HPV-16 virus-like particles (VLP16) with vaccine-induced regression of CIN III in patients immunized with this vaccine.
* Determine the efficacy of this vaccine in patients whose CIN III is associated with HPV-16 infection vs other HPV types.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 treatment groups.

All patients receive SGN-00101 subcutaneously once monthly on months 1-3 (for a total of 3 vaccinations) in the absence of disease progression or unacceptable toxicity.

* Group 1: Four months after the first vaccination, patients undergo therapeutic and diagnostic loop electrosurgical excision procedure (LEEP) or core biopsy.
* Group 2: Six months after the first vaccination, patients undergo therapeutic and diagnostic LEEP or core biopsy.

Patients in group 1 are followed at 12 months and patients in group 2 are followed at 14 months after the first vaccination.

PROJECTED ACCRUAL: A total of 66 patients (36 for group 1 and 30 for group 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade III cervical intraepithelial neoplasia (CIN III) with colposcopically visible cervical lesions
* No positive endocervical curettage or inadequate colposcopy at the time of initial cervical biopsy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm^3
* Lymphocyte count at least 500/mm^3
* Platelet count at least 150,000/mm^3
* Hemoglobin at least 10 g/dL
* No significant hematologic disease that is uncontrolled with standard therapy

Hepatic

* Bilirubin no greater than 2 mg/dL
* Liver enzymes no greater than 2.5 times normal
* No significant hepatic disease that is uncontrolled with standard therapy

Renal

* Creatinine no greater than 2 mg/dL
* No significant renal disease that is uncontrolled with standard therapy

Cardiovascular

* No significant cardiovascular disease that is uncontrolled with standard therapy

Pulmonary

* No significant respiratory disease that is uncontrolled with standard therapy
* No history of asthma

Immunologic

* HIV negative
* No clinical evidence of immunosuppression
* No autoimmune disease
* No history of allergic reactions attributed to compounds of similar chemical or biological activity as those used in this study
* No history of a positive purified protein derivative (PPD) or Tine test

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Good health based upon the results of a medical history, physical examination, vital signs, and laboratory profile
* No uncontrolled chronic disease

  * Chronic disease requiring medication is allowed provided the patient is not taking immunosuppressive drugs
* No significant endocrine (e.g., thyroid or diabetes), neurologic, gastrointestinal, or dermatologic disease that is uncontrolled with standard therapy
* No other underlying or unstable disease that would be exacerbated by the study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior BCG vaccination
* No other concurrent vaccine therapy

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* More than 30 days since prior oral or parenteral glucocorticoid steroid

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior participation in another investigational study
* No concurrent cytotoxic therapy
* No other concurrent investigational agents
* No other concurrent investigational or commercial agents or therapies intended to treat CIN

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Rate of regression | 4 months after completion of treatment
Toxicity | 4 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn D. Runowicz, MD, Study Chair — UConn Health; Mark H. Einstein, MD, MS — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York

REFERENCES:
- [Result] Einstein MH, Kadish AS, Burk RD, Kim MY, Wadler S, Streicher H, Goldberg GL, Runowicz CD. Heat shock fusion protein-based immunotherapy for treatment of cervical intraepithelial neoplasia III. Gynecol Oncol. 2007 Sep;106(3):453-60. doi: 10.1016/j.ygyno.2007.04.038. Epub 2007 Jun 22. PMID 17586030